CLINICAL TRIAL: NCT03018652
Title: Feasibility and Safety of Immunoglobulin (Ig) Treatment in COPD Outpatients With Frequent Exacerbations: Pilot Study 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IgPRx in AECOPD outpatient
Record Dates: First submitted 2016-12-16; First posted 2017-01-12 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Ig; IPRAC; outpatient
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): IVIG 0.5 g/kg, up to maximum of 80 grams will be given on the day of randomization and then every 4 ± 1 weeks for 44 weeks (Total 48 weeks) n=8
  Interventions: Drug: Intravenous immunoglobulin
- Control group (Placebo Comparator): Normal saline (0.9% NaCl) 5 mL/kg, up to maximum of 800 mL will be given on the day of randomization (this will match the volume of 0.5g/kg of IVIG product) and then every 4 ± 1 weeks for 44 weeks (Total 48 weeks) n=8
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Intravenous immunoglobulin — IVIG 0.5 g/kg, up to maximum of 80 grams will be given on the day of randomization and then every 4 ± 1 weeks for 44 weeks (Total 48 weeks)
  Arms: Intervention group
Drug: Normal Saline — 5 mL/kg, up to maximum of 800 mL will be given on the day of randomization (this will match the volume of 0.5g/kg of IVIG product) and then every 4 ± 1 weeks for 44 weeks (Total 48 weeks)
  Arms: Control group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a progressive inflammatory disease of the airways, associated with poor health status, functional disability, significant morbidity, and increased risk of death. In Ontario, COPD is the leading cause of hospital admission and readmission, and costs the health system approximately 3 billion dollars annually. Individuals with COPD experience increased 'flare-up's' (acute exacerbations) as their disease worsens, characterized by periods of increased shortness of breath, cough, phlegm production, and weakness. Acute exacerbations of COPD (AECOPD) are most commonly caused by viral or bacterial infections, and often require patients to seek attention at the emergency room or hospital for treatment. Current treatments to prevent COPD exacerbations are only modestly effective. New therapies are needed to improve the quality of life and clinical outcomes for individuals living with COPD.

Previous research at our center has shown a favourable effect of an antibody treatment (immunoglobulin) on the frequency of AECOPD, doctor visits, treatments, and hospitalizations for COPD patients. However, rigorous studies with more patients are required to confirm this effect.

The investigators propose a clinical trial to evaluate immunoglobulin treatment in outpatients with frequent exacerbations. In this study the investigators will determine if immunoglobulin treatment is feasible, safe, tolerable, and potentially effective in reducing the frequency of acute exacerbations. If this study is feasible and potentially effective, it will inform larger studies to confirm the therapeutic effect of immunoglobulin treatment, and would be a major advance in care of COPD.

DETAILED DESCRIPTION:
COPD is an incurable respiratory disease characterized by progressive decline in lung function, shortness of breath, exercise limitation, poor health status, and increased mortality. The World Health Organization cites Chronic Obstructive Pulmonary Disease (COPD) as the third leading cause of death worldwide, and estimates suggest it currently affects 65 million people. COPD is a leading cause for hospital admission and readmission in North America, and costs our health system 50 billion dollars annually.

Patients with COPD experience episodic flares of their disease, known as acute exacerbations (AECOPD). AECOPD are characterized by increased cough, shortness of breath, sputum production, weakness, and worsening airflow obstruction. There is also a high degree of systemic inflammation and immune system activation during the exacerbation. As the severity of COPD increases, the frequency of exacerbations increases as well. However, a major predictor of recurrent exacerbations is a history of exacerbation.

COPD exacerbations have a significant impact on the individual patient and the health system. Previous studies have shown that patients with exacerbations experience reductions in quality of life, such as ability to engage in activities of daily living, a worsening of lung function and an increased risk for mortality during and after the exacerbation period. Exacerbation events often cause the patient to seek acute medical attention and admission to hospital, which drives the high health care costs. History of hospital admission due to AECOPD is the strongest risk factor for readmission for recurrent AECOPD within one year. Hospitalization for AECOPD is also associated with lower 3-year survival (82.1%; 95% CI, 78.1% - 86.4%) as compared to COPD patients without history of hospitalization (92%; 95%CI, 90.8% - 93.3%) in the previous 3 years independent of the severity of airflow limitation. As a result, research has focused on methods to prevent or reduce the frequency of acute exacerbations, with expected positive impacts on patients and the health system.

Unfortunately, there is no cure for COPD, and highly effective therapies are currently lacking. The current GOLD COPD guidelines recommend smoking cessation, exercise training, maximal bronchodilator therapy, and influenza and pneumococcal vaccinations to try and prevent exacerbations. In patients with frequent exacerbations, both chronic macrolide therapy with azithromycin, N-acetylcysteine and roflumilast (a PDE-4 inhibitor) have been shown to increase the time to next exacerbation. However, these therapies are only modestly effective, and patients continue to experience exacerbations while on maximal therapy. Further research into new therapeutics to prevent and reduce exacerbations is imperative. The development of newer immunomodulatory agents as adjuvant therapy to prevent AECOPD has become an area of intense investigation.

Prolonged steroid use is associated with hypogammaglobulinemia in asthmatic patients. Patients with COPD have lower immunoglobulin G (IgG) levels compared to patients with other lung diseases, independent of oral steroid use and age. However, recurrent exacerbations still occur despite having normal baseline serum IgG (data not yet published). Intravenous and subcutaneous immunoglobulins (IVIG and SCIG, respectively) are prepared from pooled plasma from thousands of healthy blood donors. The large donor pool ensures a diversity of antibody specificities to a wide spectrum of antigens and microbial pathogens. IVIG or SCIG represents a privileged source of natural antibodies (NAb), which occur in the absence of autoimmune disease or immunization. NAb are not only an immune defense against pathogens but also have anti-inflammatory and immunomodulatory activities. Given the heightened systemic and airway inflammatory activity in patients with COPD, their propensity to infection-triggered exacerbations, and their suppressed mucosal or systemic immunity, the anti-inflammatory, anti-infective and immunomodulatory effects of Ig preparations could be beneficial for patients with COPD.

The investigators recently reported a retrospective single center self-interval analysis of Ig treatment as adjunctive preventative treatment for AECOPD in 14 patients. Half (8 patients) had at least severe COPD by GOLD criteria. Ig treatment significantly reduced moderate and severe AECOPD from 4.7 ± 3.1 to 0.6 ± 1.0 per patient-year. Number of hospitalizations was markedly reduced from twelve in the year prior to one in the year following Ig treatment initiation. Even though the median baseline IgG level in this study cohort was 5.9 g/L (interquartile range 4.1 - 7.4), and 36% had IgG less than 5 g/L, the clinical effect of Ig treatment in reducing moderate and severe AECOPD was consistent across all cases. While this demonstrates some promise, prospective controlled studies are required to determine if Ig treatment could have any impact on the frequency of COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with frequent exacerbations of COPD (clinically dominant COPD in the case of multiple co-morbidities eg. bronchiectasis, interstitial lung disease, congestive heart failure)
* Confirmed diagnosis of COPD (bronchodilator FEV1/FVC ratio <0.7 on spirometry within previous 12 months)
* Age >40 years
* >10 pack year smoking history
* Frequent COPD exacerbations in the previous 12 months before enrollment, defined by one or both of the following:
* Treatment as an outpatient with antibiotics or prednisone (physician diagnosed COPD exacerbation) on 2 previous occasions OR
* One hospitalization for COPD exacerbation (as defined by 2/3 of increased dyspnea, sputum volume, or sputum purulence in patients with known airflow limitation)
* Expected to live > 12 months

Exclusion Criteria:

* Known severe hypersensitivity to immunoglobulin or its components (anaphylaxis)
* Active or metastatic malignancy (including chronic lymphocytic leukemia) excluding local skin cancers
* History of hematopoietic stem cell transplant or solid organ transplant
* Current treatment with a biological therapy for other conditions
* Concomitant significant immunodeficiency or use of immunosuppressive treatment (other than for COPD)
* Alpha-1 antitrypsin deficiency (based on enzyme level from bloodwork)
* Significant proteinuria (dipstick proteinuria ≥ 3+ AND known urinary protein loss ≥ 2 g/day or nephrotic syndrome) and/or has a history of acute renal failure and/or severe renal impairment (creatinine more than 2.5 times the upper limit of normal and/or on dialysis)
* IgA deficiency (IgA <0.1 g/L)
* Immunoglobulin therapy in the last 12 months or on current Ig therapy or have a clinical indication for Ig replacement therapy (www.nacblood.ca/resources/guidelines/IVIG.html)
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Recruitment | 52 weeks
  Average number of patients being recruited per month. The study meets primary outcome if at least 4 patients can be recruited per month on average.
Adherence and protocol compliance | 104 weeks
  Number and percentage of recruited patients adhere to the allocated treatment and protocol. The investigators aim to achieve 80% adherence rate which is defined as at least 80% of patients adhere to 80% of allocated treatment and protocol

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | 104 weeks
  This will be assessed by documentation of adverse events in patients treated with Ig treatment versus control
Proportion of patients able to complete treatment | 104 weeks
  The proportion of patients able to complete the treatment in the experimental arm during the study period versus in the control arm
Efficacy trend: Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) rates | 104 weeks
  AECOPD will be ascertained by monthly follow-up phone calls as well as questionnaires during study visits to detect inpatient/outpatient treatment for exacerbations.
Efficacy trend: Health status | 104 weeks
  Measured by the validated St. George Respiratory Questionnaire
Efficacy trend: Quality of life | 104 weeks
  Validated quality of life measurement tool - EuroWol EQ-5D-5L
Efficacy trend: % predicted FEV1 | 104 weeks
  FEV1 value will be measured using a hand held spirometer. FEV1 value will be recorded in Litres (L) and reported as a percent of their predicted value (using the NHANES III reference standards for predicted values
Efficacy trend: FEV1/FVC | 104 weeks
  FVC will be measured using a hand held spirometer, and will be recorded in Litres (L). Ratio of FEV1 and FVC will be reported.
Efficacy trend: Health services use | 104 weeks
  Number of non-study physician visits, emergency department (ED) and hospital admissions over the twelve-month study period.
Efficacy trend: Health care system cost | 104 weeks
  Through the perspective of healthcare system, the cost of health services use and intervention will be measured. Intervention cost includes medication, staff, and equipment cost.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Cowan J, Mulpuru S, Abdallah SJ, Chopra A, Purssell A, McGuinty M, Alvarez GG, Giulivi A, Corrales-Medina V, MacFadden D, Boyle L, Hasimja D, Thavorn K, Mallick R, Aaron SD, Cameron DW. A Randomized Double-Blind Placebo-Control Feasibility Trial of Immunoglobulin Treatment for Prevention of Recurrent Acute Exacerbations of COPD. Int J Chron Obstruct Pulmon Dis. 2021 Dec 3;16:3275-3284. doi: 10.2147/COPD.S338849. eCollection 2021. PMID 34887657
- [Derived] Cowan J, Mulpuru S, Aaron S, Alvarez G, Giulivi A, Corrales-Medina V, Thiruganasambandamoorthy V, Thavorn K, Mallick R, Cameron DW. Study protocol: a randomized, double-blind, parallel, two-arm, placebo control trial investigating the feasibility and safety of immunoglobulin treatment in COPD patients for prevention of frequent recurrent exacerbations. Pilot Feasibility Stud. 2018 Aug 11;4:135. doi: 10.1186/s40814-018-0327-z. eCollection 2018. PMID 30116551